CLINICAL TRIAL: NCT05166317
Title: Comparative Efficacy of Various Non-invasive Methods in Assessing Response to Beta-blockers as Secondary Prophylaxis for Acute Variceal Bleed.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Bleed-01
Record Dates: First submitted 2021-10-08; First posted 2021-12-21 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-10

CONDITIONS: Acute Variceal Bleed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver Cirrhosis: All the consecutive patients of cirrhosis admitted to Intensive care unit of Hepatology department of ILBS.
  Interventions: Other: This is an observational study

INTERVENTIONS:
Other: This is an observational study — This is an observational study

SUMMARY:
Portal hypertension (PH) is a common complication of chronic liver disease and a major cause of morbidity and mortality in cirrhotic patients. One of the most serious complications of liver cirrhosis is esophageal varices (EV) bleeding. The hepatic venous pressure gradient (HVPG) is the gold standard for detecting portal hypertension and its complications. Furthermore, HVPG is the most reliable method for assessing the efficacy of treatment with nonselective -blockers (NSBB), which is the preferred therapy in patients with EV who are at high risk of bleeding (HRV) and as a secondary prophylaxis in the prevention of rebleed. However, the HVPG is an invasive method that is not widely used and necessitates specialized skills. For these reasons, clinical research over the last decade has been focused on identifying non-invasive tests (NITs) capable of evaluating the PH degree and its changes. The most investigated non-invasive tests are liver and splenic stiffness measurement. In advanced cirrhosis, the increase in portal pressure is less dependent on intrahepatic resistance to portal flow due to fibrosis progression and more dependent on extra-hepatic factors such as hyperdynamic circulation and splanchnic vasodilation hence correlation between LSM and PH decreases for HVPG values higher than 12 mmHg.

DETAILED DESCRIPTION:
Aim:

To determine the diagnostic accuracy of non-invasive tests in predicting response to NSBB for secondary prophylaxis of variceal bleed at 6wks.

Primary objective:

To compare the diagnostic accuracy of non-invasive modalities in correctly predicting response to beta-blockers as compared with HVPG in preventing variceal rebleed at 6 weeks.

Secondary objectives:

* Assessment of severity of portal hypertension by non-invasive methods.
* Correlation and Cut-off values for non-invasive methods in responders and non-responders.
* AAR, APRI, FIB-4 index, CSPH risk score,fibrosis index, GPR, King's score, Lok score are other non- invasive tests.
* Correlation between HVPG &non invasive test, responder and non-responder.
* Comparison ofhypersplenism(Splenic volume and area) and hematological parameters before and after treatment.
* Diagnosis and response assessment by convolutional neural network- AI based model.
* Prognostic implication of HVPG rebleed on EVL+beta-blockers.

Methodology:

* Study population:All the consecutive patients of cirrhosis admitted to Intensive care unit of Hepatology department of ILBS will be evaluated for inclusion
* Study design: Prospective observational study. The study will be conducted in Department of Hepatology ILBS.
* Study period: 1.5 years
* Sample size: Assuming that Sn of 92%, α of 5%, Power 80, we need to have 186 patients. So we decided to enroll ~200 cases (Including 5% defaulter rate)

Intervention:

* HVPG done at the baseline within 5days of acute variceal bleed and at 6weeks
* Endoscopic variceal band ligation at 3rd week
* NSBB started on day 6 which optimised according to heart rate and continued for 6 weeks.
* Monitoring and assessment
* Patients with acute variceal bleed after endovariceal band ligation will be undergoing HVPG, TE to measure splenic stiffness and baseline investigations such as complete blood count, liver and kidney function test, ultrasonography of the abdomen, contrast enhanced computerized tomography of abdomen. These investigations will be carried out within 5days. After 5 days NSBB is started and is optimsed to maximum dose according to heart rate and blood pressure. After 3 weeks EVL is done. After 6 weeks of NSBB, after 3weeks of secondary EVL;HVPG, TE to measure liver and splenic stiffness and other baseline investigations are done.

  • Hepatic venous pressure gradient (HVPG):
* Prior to the HVPG measurement, a venous access was performed under ultrasonography after local anesthesia. The Seldinger technique was used to insert a catheter into the right brachial vein or the right internal jugular vein. An occlusion balloon catheter of 6 F was guided in a branch of the hepatic veins, usually the median or right vein, under fluoroscopic control and continuous electrocardiographic and pressure monitoring.
* After inflating the balloon at the catheter's tip (maximum diameter ranges from 8.5-11.5 mm), a venous check was performed to demonstrate complete vessel occlusion. The wedged hepatic vein pressure (WHVP) was measured in this condition. Following that, the free hepatic vein pressure (FHVP) was measured after deflating the balloon at the catheter's tip. On a multi-channel recorder, a permanent trace was obtained. Pressures were also achieved in the inferior vena cava and the right atrium. According to the Baveno VI consensus, the HVPG-response was defined as a 20% or 12 mmHg reduction in HVPG after NSBB treatment.
* HVPG= WHVP - FHVP (Normal is <5mm of Hg)

  • Ultrasonography of the abdomen:
* dilated portal vein (>13 mm): non-specific
* biphasic or reverse flow in portal vein (late stage): pathognomonic
* recanalization of paraumbilical vein: pathognomonic
* portal-systemic collateral pathways (collateral vessels/varices)
* splenomegaly
* ascites
* The damping index (showing changes in the doppler hepatic vein waveform) corresponds with hemodynamically significant portal hypertension and HVPG values (together with HVPG changes after treatment)
* splenic arterial resistive index

  • Liver and splenic stiffness:
* A 3.5-MHz ultrasound transducer probe is mounted on the axis of a vibrator in the FibroScan device. Mild amplitude, low-frequency (50 Hz) vibrations are transmitted to the liver tissue, causing an elastic shear wave to propagate through the underlying tissue.If the success rate was greater than 60% and the interquartile range (IQR) was greater than 30% of the median value, LS values were accepted.
* Guidelines for measuring SS is same as LS. SS was performed on a supine patient with maximal abduction of the left arm, with the probe positioned in an intercostal space where the spleen was correctly visualized by US. Furthermore, in accordance with the FibroScan's technical features, patients with a splenic parenchymal thickness of >4 cm under the probe were excluded.

  • Radiomics:
* Convolutional neural network - Deep learning using liver and splenic channels for assessment of portal hypertension.
* STATISTICAL ANALYSIS:
* Continuous variables are expressed as the median and categorical data as numbers (percentages) (range). For group comparison, use the Mann-Whitney test for continuous variables and the 2 test for categorical variables. The Pearson correlation coefficient will be used to assess the linear relationship between noninvasive tests and HVPG (r). Receiver operating characteristic (ROC) curves will be computed for each of the diagnostic parameters evaluated (age, transaminases, platelet count, spleen diameter, Plt/Spl, LS, SS, LSPS), as well as the area under the ROC curve (AUROC).For all tests, p≤ 0.05 will be considered statistically significant. Analysis will be performed using SPSS .The analysis will be done with intention to treat and per protocol analysis if applicable.
* Adverse effects:
* 1. Major Sideeffects of Betablockers
* Bradycardia,Heart block
* Hyperglycaemia
* Heart failure
* Increase in airway resistance
* Worsening lipid profile
* Exacerbration of peripheral vascular disease

  2. HVPG related complications
* Transient arrhythmias
* Vagal reaction
* Local access pain and bleeding
* Stopping rule: Development of serious adverse effects leading to withdrawal of the drug or death from any cause.

ELIGIBILITY:
Inclusion Criteria:

* Clinical / radiological /histologic diagnosis of cirrhosis (Child A&B)
* Age >18 years
* Advanced compensated liver disease of different etiology(Viral,metabolic,alcoholic)
* Upper GI bleed
* Valid consent
* No history of NSBB use in last 6 weeks

Exclusion Criteria:

* Age > 70 years
* Portal vein thrombosis
* Underlaying shunts
* Spleen anteroposterior diameter <4cm
* Non cirrhotic portal hypertension
* Only PHG, Ectopic varices
* Heart rate <50bpm, SBP<100mm of Hg,Asthma, COPD, Aortic disease, atrioventricular block, Peripheral vascular disease.
* Pregnancy
* obese(BMI>30mm of Hg)
* HIV
* HCC / Other malignancy
* Other Comorbidities: Chronic kidney disease [ CrCl< 30] Cirrhosis : Child C Stroke Cardiac failure, Uncontrolled diabetes(HbA1c >9)
* AST/ALT >5 times
* Drug allergies
* ACLF
* Narrow intercoastal space
* Failure to give informed consent from family members.
* Patient enrolled in other clinical study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the consecutive patients of cirrhosis admitted to Intensive care unit of Hepatology department of ILBS will be evaluated for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-10 (Estimated); Primary Completion 2022-10-10 (Estimated); Study Completion 2022-10-10 (Estimated)

PRIMARY OUTCOMES:
Change in HVPG and its correlation with non-invasive methods. | 6 Weeks

SECONDARY OUTCOMES:
Assessment of severity of portal hypertension by non-invasive methods. | 6 weeks
Correlation and Cut-off values for non-invasive methods in responders and non-responders in relation to HVPG. | 6 weeks
  Non invasive methods - LSM,SSM & LSPS
Correlation of Serological and radiological non invasive tests response in comparison with HVPG. | 6 weeks
  AAR, APRI, FIB-4 index, CSPH risk score,fibrosis index, GPR, King's score, Lok score are other non- invasive tests.
Comparison of hypersplenism (Splenic volume and area) and hematological parameters before and after treatment. | 6 weeks
Diagnosis and response assessment by convolutional neural network- AI based model. | 6 weeks
Prognostic implication of HVPG rebleed on EVL+beta-blockers. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India